CLINICAL TRIAL: NCT00139347
Title: A Multi-country & Multi-center Study to Assess the Efficacy, Immunogenicity & Safety of Two Doses of GSK Biologicals' Oral Live Attenuated HRV Vaccine Given Concomitantly With Routine EPI Vaccinations Including OPV in Healthy Infants
Brief Title: Study of 2 Doses of HRV Vaccine Given Concomitantly With Routine EPI Vaccinations Including OPV in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 444563/024
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

INTERVENTIONS:
Biological: 2-dose oral live attenuated G1P[8] human rotavirus vaccine

SUMMARY:
The main objectives of this study is to determine vaccine efficacy against severe rotavirus (RV) gastroenteritis (GE) during the period starting from 2 weeks after Dose 2 until one year of age.

DETAILED DESCRIPTION:
The study has two groups: Group HRV and Group Placebo. Two oral doses administered to healthy infants who are 6-12 weeks of age at the time of Dose 1, according to a 0, 1 to 2-month schedule. Routine EPI vaccinations are given at the discretion of the investigator and according to local National Plans of Immunisation schedule in each participating country.

ELIGIBILITY:
Inclusion criteria:

* Healthy infants 6 -12 weeks old at Dose 1 with written informed consent.

Exclusion criteria:

* Allergic reaction to vaccine components;
* clinically significant history of chronic GI disease (uncorrected GI congenital malformation) or other serious medical condition per investigator, received vaccines or treatment prohibited by the protocol;
* immunocompromised.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6360
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of severe RV GE caused by the wild RV strains during the period starting from 2 weeks after Dose 2 until 1 year old.

SECONDARY OUTCOMES:
Vaccine efficacy against severe rotavirus gastroenteritis by serotypes until 1 year of age; Safety; Immunogenicity of HRV and co-administered EPI vaccines

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Argentina (8):
  - GSK Investigational Site, Colonia Caroya, Córdoba Province
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Río Cuarto, Córdoba Province
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Tunuyán, Mendoza Province
  - GSK Investigational Site, Villanueva, Mendoza Province
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, La Plata
- GSK Investigational Site, Porto Alegre, Rio Grande do Sul, Brazil
- Colombia (3):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Cali Colombia
- Dominican Republic (2):
  - GSK Investigational Site, Santo Domingo, Distrito Nacional, Sant Dom- Distrito Nacional
  - GSK Investigational Site, Santo Domingo
- GSK Investigational Site, Comayagüela, Honduras
- Panama (2):
  - GSK Investigational Site, David, Chiriquí Province
  - GSK Investigational Site, Panama City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Gonzalez Ayala et al. Co-administration with rotavirus vaccine rix4414 (rotarix™) does not interfere with the immunogenicity of oral polio vaccine (OPV). Poster presented at WSPID Bangkok, Thailand, 15-18 Nov 2007.
- [Background] Lopez P et al. Immunogenicity of an Oral Polio Vaccine is Unaffected when Co-Administered with a Human Rotavirus Vaccine RIX4414 (Rotarix™) in Latin America. Poster presented at the 13th International Congress on Infectious Diseases (ICID), Kuala Lumpur, Malaysia, 19-22 June 2008.
- [Background] Tregnaghi MW, Abate HJ, Valencia A, Lopez P, Da Silveira TR, Rivera L, Rivera Medina DM, Saez-Llorens X, Gonzalez Ayala SE, De Leon T, Van Doorn LJ, Pilar Rubio MD, Suryakiran PV, Casellas JM, Ortega-Barria E, Smolenov IV, Han HH; Rota-024 Study Group. Human rotavirus vaccine is highly efficacious when coadministered with routine expanded program of immunization vaccines including oral poliovirus vaccine in Latin America. Pediatr Infect Dis J. 2011 Jun;30(6):e103-8. doi: 10.1097/INF.0b013e3182138278. PMID 21378594
- [Background] Tregnaghi M et al. Oral Human Rotavirus Vaccine RIX4414(Rotarix™) Co-administered with Routine EPI Vaccinations Including Oral Polio Vaccine(OPV) Is Highly Efficacious in Latin-America. Poster presented at the 13th International Congress on Infectious Diseases (ICID), Kuala Lumpur, Malaysia, 19-22 June 2008.
- [Derived] Ruiz-Palacios GM, Perez-Schael I, Velazquez FR, Abate H, Breuer T, Clemens SC, Cheuvart B, Espinoza F, Gillard P, Innis BL, Cervantes Y, Linhares AC, Lopez P, Macias-Parra M, Ortega-Barria E, Richardson V, Rivera-Medina DM, Rivera L, Salinas B, Pavia-Ruz N, Salmeron J, Ruttimann R, Tinoco JC, Rubio P, Nunez E, Guerrero ML, Yarzabal JP, Damaso S, Tornieporth N, Saez-Llorens X, Vergara RF, Vesikari T, Bouckenooghe A, Clemens R, De Vos B, O'Ryan M; Human Rotavirus Vaccine Study Group. Safety and efficacy of an attenuated vaccine against severe rotavirus gastroenteritis. N Engl J Med. 2006 Jan 5;354(1):11-22. doi: 10.1056/NEJMoa052434. PMID 16394298
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 444563/024 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register